CLINICAL TRIAL: NCT06412536
Title: Triage Survey for Cardiovascular, Obesity, and Related Endocrine Trial Eligibility (SWIFT-CORE-101)
Brief Title: Triage Survey for Cardiovascular, Obesity, and Related Endocrine Trial Eligibility
Acronym: SWIFT-CORE-101
Status: Recruiting | Type: Observational
Sponsor: Brooklyn Clinical Research (Network)
Responsible Party: Sponsor
Other Study IDs: CORE042024
Record Dates: First submitted 2024-05-06; First posted 2024-05-14 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-05

CONDITIONS: Cardiovascular Diseases; Obesity; PreDiabetes; Diabetes Type 2; Metabolic Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Obesity; Prediabetic State; Diabetes Mellitus, Type 2; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Blood work — Blood work on some participants to review eligibility for future clinical trials

SUMMARY:
SWIFT-CORE-101 is a single site survey study designed to assess potential participants' eligibility to screen for industry-sponsored clinical trials. A physician will oversee the informed consent process, after which participants will be surveyed on demographics, medical history, comorbidities, and current symptoms. Site staff may collect vital signs, urine drug screens, blood draws, and urine pregnancy tests. A doctor will review medical history with the participant to determine study suitability via clinical interview. The doctor may reach out to the patient's current treating physicians and pharmacies to determine eligibility for clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Participant or Legally Authorized Representative has signed an ICF prior to study-specific procedures being performed.
2. Participant is at least 18 years old.

Exclusion Criteria:

1. Participant is pregnant, breast-feeding, or planning to become pregnant.
2. History of a clinically significant illness which in the investigator's opinion may impact participant safety or the ability to analyze study results.
3. Moderate or severe substance use disorder within 90 days prior to screen
4. Any condition that in the investigator's opinion makes a participant unsuitable for the study.
5. Currently employed by Swift Clinical Research Group, Inc. or any of its subsidiaries, including Brooklyn Clinical Research, or a first-degree relative of an employee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In year one of the program, we anticipate 4000 participants of any sex, age 18+, who have expressed interest in participating in an industry-sponsored clinical trial of an investigational product for indications in cardiovascular, obesity, and endocrine-related therapeutic areas will be screened for clinical appropriateness for a study trial.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2029-04-10 (Estimated); Study Completion 2029-04-17 (Estimated)

PRIMARY OUTCOMES:
Number of participants who are interested in industry-sponsored clinical research | 5 years
  Number of participants who are interested in industry-sponsored clinical research in each of the following therapeutic areas: cardiovascular, obesity, and endocrine.

SECONDARY OUTCOMES:
Characteristics associated with patient populations interested in clinical trials | 5 years
  Characteristics associated with patient populations interested in clinical trials stratified by demographics and therapeutic areas

CONTACTS AND LOCATIONS:
Overall Officials: Ammara Mushtaq, MD, Principal Investigator — Brooklyn Clinical Research
Locations (1):
- Brooklyn Clinical Research, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.brooklynclinicalresearch.com/

DOCUMENTS (1):
  • Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/36/NCT06412536/ICF_000.pdf